CLINICAL TRIAL: NCT06309797
Title: Evaluation of the Effects of Using an Interdental Brush Dipped in 0.2% Hyaluronic Acid Gel on Clinical Periodontal Parameters Among Patients With Periodontitis
Brief Title: Effects of Interdental Brush Dipped in 0.2% Hyaluronic Acid Gel on Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Özlem SARAÇ ATAGÜN (Other)
Responsible Party: Sponsor-Investigator, Özlem SARAÇ ATAGÜN, assistant professor, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OSATAGUN2
Record Dates: First submitted 2024-02-29; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Periodontitis
Keywords: Periodontitis; Hyaluronic Acid; Oral Hygiene
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: single-center, single-blinded, randomized controlled trial
Who Masked: Investigator
Masking Description: The investigator carrying out the measurements was not aware of which patients were assigned to the test group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (HA group) (Experimental): the test group were asked to brush their teeth, dip the interdental brush in HA gel, and use the dipped interdental brush.
  Interventions: Device: Interdental brush+HA
- Control Group (Experimental): the control group were asked to brush their teeth and use the interdental brush for oral hygiene.
  Interventions: Device: Interdental brush

INTERVENTIONS:
Device: Interdental brush+HA — interdental brushes (TePe Munhygienprodukter AB, Malmö; TePe 0.4 mm and TePe 0.6 mm) +20 mL of 0.2% HA gel (Gengigel; Ricerfarma, Milan, Italy)
  Arms: Test (HA group)
Device: Interdental brush — interdental brushes (TePe Munhygienprodukter AB, Malmö; TePe 0.4 mm and TePe 0.6 mm)
  Arms: Control Group

SUMMARY:
This study aimed to compare the effects of using an interdental brush dipped in 0.2% HA gel with those of using a regular interdental brush on clinical periodontal parameters following SRP among patients with periodontitis.

DETAILED DESCRIPTION:
The additional use of agents with antibacterial and anti-inflammatory activities such as hyaluronic acid (HA) in treating periodontal disease has recently become popular. This study aimed to evaluate the effects of using an interdental brush dipped in 0.2% HA gel on clinical periodontal parameters.This randomized controlled trial was conducted among 33 female patients and 27 male patients with stage II/III grade A/B periodontitis. After the initial periodontal treatment, patients were randomly divided into two groups; those in the test group were asked to use an interdental brush dipped in 0.2% HA gel twice a day after brushing, while those in the control group were asked to use a regular interdental brush. Clinical periodontal parameters including the pocket depth, clinical attachment loss, gingival index, plaque index, and papillary bleeding index (PBI) were assessed at baseline and in the 1st and 3rd months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18-55 years of age
2. Being systemically healthy
3. Having periodontitis (Stage 3)
4. Not to have used any medication in the last three months
5. Not smoking
6. Right-handed
7. At least 20 natural teeth

Exclusion Criteria:

1. Patients with interdental caries
2. Patients with orthodontic appliances
3. Patients with removable (partial) prostheses
4. Patients with oral and/or peri-oral pain
5. Patients with significant oral lesions
6. Patients with antibiotic use in the last 3 months, pregnancy and breastfeeding
7. Patients who have undergone periodontal treatment within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Gingival index (GI) | Baseline-4 weeks-12 weeks
  Improvement in GI; lower scores mean a better outcome; Minimum score:0 Max.score: 3
Plaque index (PI) | Baseline-4 weeks-12 weeks
  Improvement in PI; lower scores mean a better outcome; Minimum score:0 Max.score: 5
Papillary bleeding index (PBI) | Baseline-4 weeks-12 weeks
  Improvement in PBI; lower scores mean a better outcome; Minimum score:0 Max.score: 3
Pocket depth (PD) | Baseline-4 weeks-12 weeks
  Improvement in PD; lower scores mean a better outcome
Clinical attachment loss (CAL) | Baseline-4 weeks-12 weeks
  Improvement in CAL; lower scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: özlem saraç atagün, PhD, Principal Investigator — Sağlık Bilimleri Üniversitesi Gülhane Diş Hekimliği Fakültesi Periodontoloji AD
Locations (1):
- Sağlık Bilimleri Üniversitesi Gülhane Diş Hekimliği Fakültesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarac Atagun O, Ceylan Sen S, Ustaoglu G, Ozcan E. Evaluation of the effects of using an interdental brush dipped in 0.2% hyaluronic acid gel on clinical periodontal parameters among patients with periodontitis: a randomized controlled trial. BMC Oral Health. 2025 Apr 25;25(1):635. doi: 10.1186/s12903-025-06038-7. PMID 40281514